CLINICAL TRIAL: NCT03987724
Title: The Effects of Acute Exercise on Tumor Blood Flow
Brief Title: Exercise and Tumor Blood Flow
Acronym: EXETUMOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Ilkka Heinonen, Adjunct professor, University of Turku
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: T187/2019
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Tumor Blood Flow at Rest and During Exercise
Keywords: Clinical trial; Positron emission tomography; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Intervention Model Description: Each subject will serve as their own control (tumor blood flow at rest vs. blood flow during exercise).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): The experiment consists of a supine bicycle exercise in a positron emission tomography (PET) scanner. Each subject will perform the experiment as well as serve as their own control (tumor blood flow at rest vs. blood flow during exercise).
  Interventions: Other: Positron emission tomography (PET) imaging at rest and during supine bicycle exercise

INTERVENTIONS:
Other: Positron emission tomography (PET) imaging at rest and during supine bicycle exercise — Tumor blood flow and its heterogeneity will be measured with PET at rest and during supine bicycle exercise.

SUMMARY:
This research aims at investigating tumor blood flow response to acute exercise in human cancer patients. It is hypothesized and expected that acute exercise increases tumor blood flow, which could plausibly increase the efficacy of cancer treatment.

DETAILED DESCRIPTION:
Physical activity has been applied as an adjunctive therapy in the secondary prevention of many cancers, but very little is currently known clinically and mechanistically about the effects of physical activity and exercise on tumor itself. Based on recent evidence from pre-clinical studies, it is plausible to expect that changes in tumor blood flow and its heterogeneity, oxygenation, and metabolism due to exercise would increase the delivery of chemotherapy and other cancer drugs into the tumor increasing the efficacy of cancer treatment.

Eight (8) newly diagnosed Hodgkin lymphoma cancer patients will be recruited to investigate whether these pre-clinical findings can be extended to humans to serve as an evidence-based proof-of-concept for the possible inclusion of exercise in the treatment of cancer during chemotherapy. To study the effect of acute physical exercise on tumor blood flow and its heterogeneity, supine bicycle exercise in a positron emission tomography (PET) scanner will be used to exercise Hodgkin lymphoma cancer patients. These experiments are additional measurements to their normal treatments, and no new interventional approaches will be conducted in this study.

The study consists of one fitness test assessment, and tumor blood flow measurements with PET at rest and during supine cycling exercise.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed Hodgkin lymphoma

Exclusion Criteria:

* abnormal fatigue, anemia, or physical dysfunction due to the disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-09-17 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Tumor blood flow | Tumor blood flow is measured at one time point, at least two (2) days apart from baseline fitness test assessment. Tumor blood flow at rest and during supine cycling exercise will be measured on the same day.
  Measured with PET and radiowater ([(15)O]H2O) tracer. Tumor perfusion will be determined as mean tumor blood flow.

SECONDARY OUTCOMES:
Spatial dispersion (heterogeneity) of tumor blood flow | The heterogeneity of tumor blood flow is measured at one time point, at least two (2) days apart from baseline fitness test assessment. The heterogeneity of tumor blood flow at rest and during supine cycling exercise will be measured on the same day.
  Measured with PET and radiowater ([(15)O]H2O) tracer. Tumor blood flow heterogeneity will be determined as voxel variation in perfusion divided by the mean perfusion of the voxels.

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Heinonen, PhD, Principal Investigator — University of Turku
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No